CLINICAL TRIAL: NCT01917175
Title: Research Platform " Early Identification and Treatment of Early HIV Infection in Côte d'Ivoire "
Brief Title: Early Identification and Treatment of Early HIV Infection in Côte d'Ivoire
Acronym: PRECO-CI
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS 1220/12277 PRECO-CI
Record Dates: First submitted 2013-08-05; First posted 2013-08-06 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: HIV Infection
Keywords: HIV; Cohort; Early HIV infection; Côte d'Ivoire; Disease progression
MeSH Terms: conditions — HIV Infections; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and whole blood for PBMC preparation
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV+ patients with an estimated date of seroconversion: It was estimated that 564 individuals, will be enrolled at the Blood Bank Medical Centre, including 364 individuals already followed-up (former PRIMOCI ANRS 1220 cohort started in 1997) and 200 newly enrolled individuals in this study.

SUMMARY:
Set-up of a biobank for patients with an estimated date of infection seroconverters: store plasma and cells samples at initial contact and during follow-up for future analysis and analysis in international collaborative cohort seroconverters.

ELIGIBILITY:
Inclusion Criteria:

* patients included in the last Primo-CI ANRS 1220 protocol
* All HIV infected individuals diagnosed during a blood donation with an estimated date of HIV seroconversion that will respect the following criteria: (i) age ≥18 (ii) HIV-1 or HIV-1+2 infected, (iii) HIV-seronegative at the preceding donation; (iv) who returned to the clinic to be informed of their HIV test result (v) with an HIV serology confirmed with two specific tests in two different laboratories (vi) who have never received ART for curative purpose
* informed on study objectives and have a signed informed consent.

Exclusion Criteria:

* Patient living outside of Abidjan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All HIV infected individuals that will have had a contact with the Blood Bank Medical Center since 1992.
Sampling Method: Non-Probability Sample
Enrollment: 511 (Actual)
Dates: Start 1997-06 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Natural history of HIV infection in Sub-Saharan Africa | 12 months after ART initiation
  Plasmatic HIV viral load and CD4 measured every six months and incidence of morbidity events associated with AIDS

SECONDARY OUTCOMES:
Estimate the probability of disease progression after HIV seroconversion | 12 months after ART initiation
  Disease progression will be estimated with CD4 cell loss and time from seroconversion to clinical AIDS, death and antiretroviral therapy initiation
Evolution of markers of HIV infection and immunity | 12 months after ART initiation
  CD4 count, immune activation, plasma HIV-RNA intracellular, HIV-DNA
Viral genetic diversity description | Inclusion (J0)
  biomolecular analysis of HIV-1
Primary resistance to antiretroviral treatment | Inclusion (J0)
  Frequency of primary resistance to antiretroviral treatment (genotyping)
Metabolic and lipodystrophic disorders | 12 months after ART initiation
  Metabolic analysis (Total Cholesterol, HDL and LDL, Triglycerides) and lipodystrophia measurements
Incidence of pregnancies | 12 months after ART initiation
  Occurence of pregnancies
T lymphocytes activation and evolution in seroconverters | Inclusion
  Define parameters of activation of T lymphocytes and their evolution since primo-infection among individuals recently infected in West Africa; Expression of markers CD38, HLA-DR, CD28 and CD127 on CD4 and CD8 T cells by flux cytometry
T lymphocytes activation and evolution in seroconverters | 12 months after ART initiation
  Define parameters of activation of T lymphocytes and their evolution since primo-infection among individuals recently infected in West Africa; Expression of markers CD38, HLA-DR, CD28 and CD127 on CD4 and CD8 T cells by flux cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Albert Kla Minga, MD, PhD, Principal Investigator — CMSDS, Abidjan, Côte d'Ivoire; Patrick Coffie, MD, PhD, Principal Investigator — Programme PACCI, Abidjan, Côte d'Ivoire; Charlotte Lewden, MD, PhD, Principal Investigator — Institut de Santé Publique, d'Epidémiologie et de Développement (ISPED), Bordeaux, France
Locations (2):
- Côte d’Ivoire (2):
  - Centre Médical du Suivi des Donneurs de Sang (Blood Bank Medical Centre), Abidjan
  - Centre National de Transfusion Sanguine (National Blood Transfusion Centre), Abidjan

REFERENCES:
- See also: Sponsor site — http://anrs.fr/
- See also: Methodology centre site — http://mereva.net